CLINICAL TRIAL: NCT03846076
Title: Investigating Treatment and Information Processing in Olfactory Reference Syndrome: A Pilot Study
Brief Title: Internet Delivered CBT for Olfactory Reference Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Volen Ivanov (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Sponsor-Investigator, Volen Ivanov, Principal Investigator, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-00775
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2021-11-02 (Actual); Status verified 2021-11

CONDITIONS: Olfactory Reference Syndrome
MeSH Terms: conditions — olfactory reference syndrome | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-delivered CBT (Experimental): 10 weeks of CBT delivered via the Internet.
  Interventions: Behavioral: Cognitive behavioral therapy

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy — Cognitive behavioral therapy

SUMMARY:
The primary aim of the study is to test the feasibility and efficacy of, a manual based, Internet-delivered, cognitive behaviour therapy (CBT) for patients with Olfactory Reference Syndrome (ORS) who live in Sweden. The secondary aim is to investigate smell sensitivity and body odor in these ORS-patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of ORS
* Outpatients
* Male or female
* Signed informed consent
* Have regular access to a computer with Internet access and skills to use the web

Exclusion Criteria:

* Not able to read or understand the basics of the ICBT self-help material
* Psychotropic medication changes within two months prior to treatment
* Completed CBT for ORS within last 12 months
* Ongoing substance dependence or misuse
* Lifetime bipolar disorder or psychosis
* Suicidal ideation
* Axis II diagnosis that could jeopardize treatment participation
* Serious physical illness that will be an obstacle in ICBT
* Other ongoing psychological treatments that could affect ORS symptoms
* Epilepsia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for olfactory reference syndrome (ORS-YBOCS) | Change from baseline (week 0) to post-treatment (week 10).
  The instrument is a 12-item clinician-administered scale rating the severity of ORS symptoms during the past week. Each item is scored along a Likert scale ranging from 0 (least extreme) to 4 (most extreme), with higher total scores indicating more severe ORS symptoms (range 0-48).

SECONDARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for olfactory reference syndrome - Self Report (ORS-YBOCS-SR) | Change from baseline (week 0) to post-treatment (week 10).
  The instrument is a12-item self-administered scale rating the severity of ORS symptoms during the past week.
  Each item is scored along a Likert scale ranging from 0 (least extreme) to 4 (most extreme), with higher total scores indicating more severe ORS symptoms (range 0-48).
The Montgomery Åsberg Depression Rating Scale - self report (MADRS-S) | Change from baseline (week 0) to post-treatment (week 10).

CONTACTS AND LOCATIONS:
Locations (1):
- M46: Karolinska Universitetssjukhuset, Psykiatri Sydväst Stockholm, Huddinge, Sweden, 141 86, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided